CLINICAL TRIAL: NCT06814171
Title: Long-term Impact of a Low-carbohydrate Versus Low-fat Breakfast on Blood Glucose Control in Type 2 Diabetes
Brief Title: UBC Breakfast Study 2.0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Dr., University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H25-00043
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate breakfast (Experimental)
  Interventions: Other: Low-carbohydrate breakfast
- Low-fat Control breakfast (Active Comparator)
  Interventions: Other: Low-fat Control breakfast

INTERVENTIONS:
Other: Low-carbohydrate breakfast — Daily low-carbohydrate breakfasts for one year.
  Arms: Low-carbohydrate breakfast
Other: Low-fat Control breakfast — Low-fat breakfasts for one year.
  Arms: Low-fat Control breakfast

SUMMARY:
Type 2 diabetes (T2D), a prevalent metabolic disorder impacting >3 million Canadians, is characterized by insulin resistance and high blood glucose. Chronically elevated blood glucose (i.e., hyperglycemia) and swings in glucose (i.e., glucose variability) contribute to complications of T2D. Specifically, post-meal hyperglycemic spikes are independent risk factors for cardiovascular disease and mortality. People with T2D often exhibit a different circadian pattern from healthy individuals, with higher glucose excursions in the morning, after breakfast. This makes breakfast a crucial meal in achieving glycemic control. One strategy to reduce or eliminate this high glucose excursion is to consume a low-carbohydrate breakfast. Our recently published 3-month clinical trial (Oliveira et al., AJCN 2023) - funded by the Egg Farmers of Canada (EFC) & Egg Nutrition Center (ENC) - highlighted the positive impact of a simple dietary intervention, where individuals were advised to consume an egg-based, low-carbohydrate breakfast. This intervention led to improved glycemic control assessed by continuous glucose monitoring and reduced overall energy and carbohydrate intake when compared to a low-fat guideline breakfast. While we saw a within-group reduction HbA1c in the egg-based low-carbohydrate breakfast group, the between group difference did not reach statistical significance. Since HbA1c reflects the average glucose over the preceding 3 months, likely, our previous study's duration was not long enough to demonstrate significant reductions in HbA1c. For a low-carbohydrate breakfast to be recognized as an evidence-based strategy in nutrition and clinical practice guidelines, a longer-term study that demonstrates reductions in HbA1c is needed.

Collectively, our promising early results demonstrate that the time is right and that our team is poised to deliver a longer, well-powered randomized controlled trial (RCT) to solidify low-carbohydrate breakfasts as an evidence-based strategy to improve glucose control and improve health outcomes for people living with T2D.

DETAILED DESCRIPTION:
Research Question: Does the advice and guidance to consume a long-term low-carbohydrate breakfast impact blood glucose levels in people with type 2 diabetes?

Objectives

The specific aims are to conduct a RCT to determine if advice and guidance to consume a low-carbohydrate breakfast, compared to standard guidelines control breakfast, for one year:

Improves glycemic control assessed by HbA1c (primary outcome) in individuals with type 2 diabetes (T2D); Improves glycemic variability and lowers postprandial hyperglycemia in individuals with T2D; Reduces body weight and fat mass in individuals with T2D; Reduces feelings of hunger and consequently lowers daily energy and carbohydrate intake in individuals with T2D.

Hypothesis:

Advice and guidance to consume a low-carb high-fat breakfast, compared to a standard control low-fat breakfast over 1 year will reduce HbA1c levels; When compared to a low-fat breakfast, low-carb high-fat breakfast will improve glucose monitoring metrics.

Compared to a low-fat breakfast, a low-carb high-fat breakfast will lower feelings of self-reported hunger; A low-carb high-fat breakfast will improve body composition in individuals with T2D.

Background Information

In the years leading up the pandemic (2016 to 2019), almost 1 in 10 Canadian adults aged 20 to 79 (9%) had diabetes. The prevalence of diabetes ranged from 1% of Canadians aged 20 to 39 to almost one in five seniors aged 60 to 79 (18%) (Statistics Canada). The high prevalence is associated with a high personal, clinical and economic burden, with diabetes resulting in approximately 15,700 deaths each year in Canada (Cho et al., 2018). Clearly, strategies to improve glucose control and reduce the burden of T2D are attractive from a quality of life and economic standpoint.

Lowering dietary carbohydrate intake has been shown to improve blood glucose control and is now recognized as an evidence-based nutritional strategy in T2D (Churuangsuk et al., 2020). However, low-carbohydrate diets are often criticized as being too difficult to sustain in the long-term. One potential strategy is to limit carbohydrate intake at only one daily meal. Since the largest hyperglycemic spike usually occurs in the morning after the first meal, manipulating the carbohydrate content of the breakfast may be a simple strategy to improve glycemic control in people with T2D.[ Long-term trials specifically examining low-carbohydrate egg-based breakfasts are lacking. To our knowledge, our last RCT (Oliveira et al., AJCN 2023) is the most recent and robust evidence examining the effects of a low-carbohydrate breakfast on glucose control in T2D up to now (described in detail below). Pedersen et al. (2016) demonstrated in T2D patients that excluding carbohydrates from the first meal of the day could mitigate the significant glucose spike typically observed after breakfast. Similarly, Park et al. (2014) found that a high-protein breakfast reduced postprandial glucose concentrations without exacerbating the glucose response to subsequent meals, suggesting that incorporating more protein into breakfast could be a therapeutic approach for T2D management.

Considering our publications demonstrating enhanced glycemic control in T2D patients following a low-carbohydrate breakfast (Chang et al., 2019 and Oliveira et al., AJCN 2023), alongside existing research indicating the health benefits of "bigger" and high-protein breakfasts in T2D, there is compelling justification for conducting a longer-term, well-designed, adequately powered randomized controlled trial (RCT). We hypothesize that consuming a low-carbohydrate breakfast for 1-year will improve blood glucose control and be recognized as a scientifically substantiated, evidence-based nutritional strategy for T2D, with promise for potential incorporation into clinical practice guidelines.

Research Method

Overview

Two-hundred eighty (N=280) individuals with diagnosed T2D (30-79 years old), will be recruited from across Canada for a 1-year parallel-group remotely-delivered RCT through online and newspaper advertising, emails, third-part recruitment agency as well as word of mouth. Participants will be randomized to consume a low-carbohydrate breakfast (LC, n=140) or a low-fat "standard care" control breakfast (CTL, n=140) for 12 months, stratified by age (30-50, 51-79) and biological sex (M/F).

Participants will continue to take any medications as instructed by their physicians throughout this real-world trial but will be asked to report any changes that occur to study personnel over the 1-year period.

Experimental conditions

A 1-year parallel-group RCT is proposed. Due to the nature of the dietary intervention trial, study participants and investigators will not be blinded - however, masking will be implemented wherever possible (e.g., for data analysis). Eligible participants will be randomized to either the:

i) Low Carbohydrate Breakfast (LC, n=140) or ii) Low-fat "standard care" Control Breakfast (CTL, n=140) Both breakfasts will be consumed daily for a period of 1-year.

Breakfast options Similar to our previous trial, each group will be provided with an initial menu of 12 recipes consisting of ~400-500 kcal from which to choose each morning. LC breakfasts will contain <10% carbohydrates, 60-75% fat, and 15-30% protein (e.g., omelette with cheese) and CTL breakfasts will contain 45-70% carbohydrates, 20-40% fat, 15-25% protein (e.g., oatmeal with berries). Participants will be instructed to have their first meal of the day (before 12pm) as per recipes and to upload a daily photo of their breakfast to confirm compliance. As in our previous low-carbohydrate breakfast study no instructions will be provided for other meals as the goal is to be free-living with minimal intervention and increased potential for implementation and translation to real-world life.

Dietary intake assessment Participants will be guided to register three 3-day food records (2 weekdays and 1 weekend day) at baseline, 3, 6, 9 and 12 months of the trial through REDCap-UBC links. Macronutrient composition and total caloric intake will be calculated using ESHA software to determine any group differences across time.

Hunger and Fullness questionnaire Participants will complete a 100 mm Visual Analog Scales (VAS) to measure self-reported hunger, fullness and desire for sweet and savoury foods at multiple timepoints across one day at baseline, 3, 6, 9 and 12 months. They will be advised to fill out the survey after breakfast.

GODIN Leisure-Time Exercise Questionnaire Participants will be asked to report changes to their physical activity by completing a GODIN questionnaire through a REDCap-UBC link sent by email at baseline and end of the trial. The Godin Leisure-Time Exercise Questionnaire allows the assessment of self---reported leisure---time physical activity.

Chronotype survey (exploratory outcome) Chronotype will be determined using the Morningness-Eveningness questionnaire (MEQ) send through a REDCap-UBC link by email at baseline.

Blood testing Blood samples will be collected at baseline and after 12 months for HbA1c and lipids (triglycerides, total, HDL, and LDL cholesterol) at the nearest local laboratory with lab requisition provided by research team.

Anthropometry Anthropometric measures (height, body weight, and waist circumference) will be assessed at baseline, 3, 6, 9 and, 12 months during Zoom calls with the dietitian.

Glucose monitoring Participants in both groups will receive a flash glucose monitoring sensor (FreeStyle Libre 2) at baseline, to record their glucose levels for 14 days before starting the breakfast recipes. Once intervention has started, they will wear the flash glucose monitoring sensor for 14 days at 6 and 12 months to capture changes related to dietary approach. The sensor will be an informative tool for glycemic control in both groups by measuring daily postprandial hyperglycemia and providing the data necessary to calculate 24-hour average, post-meal incremental areas under the curve (iAUC), and glycemic variability.

ELIGIBILITY:
Inclusion Criteria:

i) physician-diagnosed T2D, ii) 30-79 years old and iii) on stable medication for at least 3 months

Exclusion Criteria:

i) Use of exogenous insulin; ii) taking more than 3 glucose lowering medications; iii) ongoing medical treatment for diseases such as cancer, auto-immune or inflammatory disease, or kidney disorders; iv) allergy, intolerance or aversion to eggs or any other dietary restrictions (e.g., vegan, breakfast skipping) that will prevent them from following the standardized study diets; v) being unable to follow the controlled diet instructions; vi) currently following a low-carbohydrate or very low-carbohydrate diet (ketogenic diet); vii) currently pregnant or lactating, or planning on becoming pregnant within the next 12 months; viii) with scheduled surgery or medical intervention that prevents following study diet; and ix) being unable to follow remote guidance by internet or smartphone.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | At baseline and after 12 months
  Blood HbA1c

SECONDARY OUTCOMES:
24 h average glucose by continuous glucose monitoring | Baseline, 6 and 12 months
  Continuous glucose monitoring for 14 days to assess 24hour average glucose
Post-meal areas under the curve [AUC] glucose by continuous glucose monitoring | Baseline, 6 and 12 months
  14 day continuous glucose monitoring to assess Post-meal areas under the curve [AUC] glucose
Glycemic variability by continuous glucose monitoring | Baseline, 6 and 12 months
  14-day continuous glucose monitoring to assess glycemic variability
Body weight | Baseline, 3, 6, 9 and, 12 months
  Self-reported body weight in kg
Body mass index | Baseline, 3, 6, 9 and, 12 months
  Calculated body mass index (BMI) as kg/m2.
Waist circumference | Baseline, 3, 6, 9 and, 12 months
  Self-measured and self reported waist circumference in inches
Triglycerides | Baseline and 12 months
  Blood triglycerides
Total cholesterol | Baseline and 12 months
  Blood total cholesterol
HDL cholesterol | Baseline and 12 months
  Blood HDL cholesterol
LDL cholesterol | Baseline and 12 months
  Blood LDL cholesterol
Energy intake | Baseline, 3, 6, 9, and 12 months
  Daily energy intake (kcal) measured by 3-day food records
Carbohydrate intake | Baseline, 3, 6, 9, and 12 months
  Daily carbohydrate intake (g) and (kcal) measured by 3-day food records
HbA1c at 6 months | 6 months
  HbA1c at 6 month

OTHER OUTCOMES:
Chronotype | Baseline
  Chronotype assessed by the Morningness-Eveningness questionnaire (MEQ)

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia - Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Compiled data will be provided upon reasonable request.

REFERENCES:
- [Background] Oliveira BF, Chang CR, Oetsch K, Falkenhain K, Crampton K, Stork M, Hoonjan M, Elliott T, Francois ME, Little JP. Impact of a Low-Carbohydrate Compared with Low-Fat Breakfast on Blood Glucose Control in Type 2 Diabetes: A Randomized Trial. Am J Clin Nutr. 2023 Jul;118(1):209-217. doi: 10.1016/j.ajcnut.2023.04.032. Epub 2023 May 29. PMID 37257563